CLINICAL TRIAL: NCT05102045
Title: The Effects of Repetitive Transcranial Magnetic Stimulation and Aerobic Exercise on Cognition, Balance and Functional Brain Networks in Patients With Alzheimer's Disease
Brief Title: The Effects of Repetitive Transcranial Magnetic Stimulation in Patients With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Miray Budak, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alzheimer.rTMS.fMRI
Record Dates: First submitted 2021-08-03; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Repetitive Transcranial Magnetic Stimulation; Cognitive Function; Aerobic Exercise; Functional MRI; Resting State Networks
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation; Exercise; Cholinesterase Inhibitors; Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TMS group (Experimental): In the TMS group (n=10) rTMS was applied to the bilateral dorsolateral prefrontal cortex (DLPFC) at 20 Hz, for 5 consecutive days per week for over 2 weeks (totally 10 sessions) in addition to the pharmacological treatment.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Drug: Acetylcholinesterase Inhibitors; Drug: Memantine
- AE group (Experimental): AE group (n=9) received a moderate- intensity aerobic exercise program lasting 50 minutes per session, 5 consecutive days per week for over 2 weeks (totally 10 sessions) in addition to the pharmacological treatment.
  Interventions: Other: Aerobic Exercise; Drug: Acetylcholinesterase Inhibitors; Drug: Memantine
- Control group (Active Comparator): No additional intervention was given to the patients in the control group (n=8) and participants were only treated pharmacologically.
  Interventions: Drug: Acetylcholinesterase Inhibitors; Drug: Memantine

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — TMS is a non-invasive application that induces changes in neuronal polarization and activity by causing the induction of weak electric currents in a rapidly changing magnetic field. Repetitive TMS (rTMS) refers to the application of regular TMS pulses at fixed intervals.
  Arms: TMS group
Other: Aerobic Exercise — Brisk exercise that promotes the circulation of oxygen through the blood and is associated with an increased rate of breathing.
  Arms: AE group
Drug: Acetylcholinesterase Inhibitors — Donepezil, Rivastigmine, Galantamine were given in combination for Alzheimer's disease.
Drug: Memantine — Memantine were given for Alzheimer's disease. .

SUMMARY:
Objectives: The purpose of this study was to investigate the effects of high-frequency repetitive Transcranial Magnetic Stimulation (rTMS) in Alzheimer's Disease (AD).

Methods: Twenty-seven AD patients aged ≥60 years were included in the study and divided into 3 groups (rTMS, Aerobic Exercise (AE) and control). All groups received pharmacological treatment. rTMS group (n=10) received 20 Hz rTMS treatment on bilateral dorsolateral prefrontal cortex, 5 days a week over 2 weeks, and AE group (n=10) received the moderate-intensity aerobic exercise for 50 min sessions, 5 days a week over 2 weeks. Control group (n=10) was only treated pharmacologically. Neuropsychiatric and behavioral status, cognition, balance, functional mobility, and quality of life, and functional brain changes were evaluated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* having clinical AD diagnosis according to the NINCDS-ADRDA (National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association) criteria
* being 60 years and older
* having Clinical Dementia Rating Scale (CDR) scores 1 or 2
* living independently

Exclusion Criteria:

* not being able to walk independently,
* having physical disabilities,
* having a history of alcohol / substance abuse,
* having head trauma
* having epileptic seizures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging | 4 weeks after baseline
  Resting state networks and activation areas in the brain were evaluating with Functional Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Neuropsychometric test battery | 4 weeks after baseline
  Neuropsychometric status was evaluated with Neuropsychometric test battery. Higher score means better result.
Mini Mental State Examination Test | 4 weeks after baseline
  General cognition was evaluated with Mini Mental State Examination Test. The functions of the individual, which are gathered under five basic headings as orientation, recording memory, attention, calculation, recall and language, are evaluated over 30 points. Higher score means better result.
Neuropsychiatric Inventory Questionnaire | 4 weeks after baseline
  Neuropsychiatric status was evaluated with The Neuropsychiatric Inventory Questionnaire.
  A total of 12 behavioral domain screening questions, including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/apathy, disinhibition, irritability/lability, abnormal motor behavior, sleep/night behaviors, appetite and eating changes. questioned according to the presence of symptoms. Otherwise, the next area is passed, and if there is, it is detailed with more specific questions related to that area. Multiplying the scores of the frequency and severity of the symptom creates the total score of that item. Higher score means worse result.
Berg Balance Scale | 4 weeks after baseline
  Balance was evaluated with Berg Balance Scale. It consists of 14 questions that evaluate whether the tasks related to balance can be fulfilled in a spectrum ranging from sitting position to standing up and standing on one leg. It is scored as 0: unable to do, 4: doing independently. The total score is 56. A fall risk of 0-20 is considered high, a fall risk of 21-40 is considered moderate, and a fall risk of 41-56 is low. Changes of 8 points or more are considered significant in terms of addiction status.Higher score means better result.
Timed Up and Go Test | 4 weeks after baseline
  Functional mobility was evaluated with Timed Up and Go Test. Time is started as soon as the person gets up from the chair and ends when he/she sits on the chair after walking 3 meters and turning. The fact that the person's walking speed is higher than the upper limit of the value range determined for the age group is associated with impaired performance. Higher score means better result.
Quality of Life in Alzheimer's Disease Scale | 4 weeks after baseline
  Quality of life was evaluated with Quality of Life in Alzheimer's Disease Measure.
  Each of the 13 items in the scale is scored on a four-point scale ranging from 1 (very poor) to 4 (excellent). The total score is between 13-52. Higher score means better result.
Frontal Behavioral Inventory | 4 weeks after baseline
  Behavioral status was evaluated with The Frontal Behavioral Inventory. It consists of 24 items including behavior and personality traits. Scoring of the scale; 0 = absent, 1 = mild / rare, 2 = moderate, 3 = severe / most of the time. The total score ranges from 0 to 72. Higher score means worse result.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budak M, Bayraktaroglu Z, Hanoglu L. The effects of repetitive transcranial magnetic stimulation and aerobic exercise on cognition, balance and functional brain networks in patients with Alzheimer's disease. Cogn Neurodyn. 2023 Feb;17(1):39-61. doi: 10.1007/s11571-022-09818-x. Epub 2022 May 30. PMID 36704634